CLINICAL TRIAL: NCT02675517
Title: Assessment of Physical Functioning and Handling of Spiolto® Respimat® in Patients With Chronic Obstructive Pulmonary Disease (COPD) Requiring Long-acting Dual Bronchodilation in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237.42
Record Dates: First submitted 2016-01-29; First posted 2016-02-05 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Spiolto Respimat: COPD patients requiring a fixed combination therapy of two long-acting bronchodilators (LAMA + LABA) according to approved Summary of Product Characteristics (SmPC) and Global Initiative for Chronic Obstructive Lung Disease (GOLD)guidelines
  Interventions: Drug: Spiolto Respimat

INTERVENTIONS:
Drug: Spiolto Respimat — Tiotropium bromide + Olodaterol

SUMMARY:
The primary objective of the study is to measure changes in physical functioning - serving as a surrogate for physical activity and exercise capacity - in COPD patients being treated with Spiolto® Respimat® after approximately 6 weeks. A secondary objective is to evaluate the patient¿s general condition (physician¿s evaluation) at visit 1 (baseline visit at the start of the study) and at visit 2 (final visit at the end of the study, approx. 6 weeks after visit 1), as well as patient satisfaction with Spiolto® Respimat® at visit 2.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent prior to participation
2. Female and male patients = 40 years of age
3. Patients diagnosed with COPD and requiring long-acting dual bronchodilation (LAMA + LABA) treatment according to approved Spiolto® Respimat® SmPC and COPD GOLD guideline recommendation

Exclusion criteria:

1. Patients with contraindications according to Spiolto® Respimat® SmPC
2. Patients who have been treated with a LABA/LAMA combination (free and fixed dose) in the previous 6 months
3. Patients continuing LABA- Inhalative Corticosteroides (iCS)treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists
4. Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks
5. Pregnancy and lactation
6. Patients currently listed for lung transplantation
7. Current participation in any clinical trial or any other non-interventional study of a drug or device

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 1737 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Germany

REFERENCES:
- [Derived] Taube C, Bayer V, Zehendner CM, Valipour A. Assessment of Patient Experiences with Respimat(R) in Everyday Clinical Practice. Pulm Ther. 2020 Dec;6(2):371-380. doi: 10.1007/s41030-020-00127-4. Epub 2020 Aug 28. PMID 32857327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1737 patients were treated. Of these 1578 patients had both visits documented as well as filled in all questionnaires, thus being evaluable for analysis of primary and secondary endpoints .
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be entered to trial drug if any of the specific entry criteria was violated.
Groups:
- Spiolto Respimat: COPD patients were administered 2.5 microgram/2.5 microgram per puff inhalation solution of the fixed combination therapy of two long-acting bronchodilators (Long-acting muscarinic antagonist (LAMA) + Long-acting beta2 adrenoceptor agonist (LABA)) via one device Respimat® for approximately 6 weeks according to approved Summary of Product Characteristics (SmPC) and the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines
Period: Overall Study
Arm/Group | Spiolto Respimat
Started | 1737
Completed | 1578
Not Completed | 159
Not completed — No evaluable PF-10 questionnaire at all | 8
Not completed — Evaluable PF-10 questionnaire at visit1 | 151

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients who had given their written informed consent to study participation, had been registered and had received at least one dose of Spiolto® Respimat® were included in the Treatet set (TS).
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 1737
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of registration was captured Population: Treated set
  Years | 66.51 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 747
  Male | 990
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Therapeutic Success at Week 6 (Approx.) (Visit 2).
Description: Therapeutic success defined as a minimum 10-point increase of Physical functioning questionnaire (PF-10 ) score after approximately 6 weeks of Spiolto® Respimat® treatment The PF-10 used for assessing the primary outcome "physical functioning" is a sub-domain of the validated Short Form 36 (SF-36) quality of life questionnaire and consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. The total score ranges from 0 to 100. A higher score indicates a better physical functioning.
Time Frame: after approximately 6 weeks
Population: Full analysis set (FAS): This analysis set consist of all screened patients with informed consent, date of registration, at least one documented administration of Spiolto® Respimat® & available PF-10 score at visit 1&2, & confirmed main diagnosis of COPD in whom treatment with long-acting anticholinergics plus bronchodilators is indicated.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 1578
Percentage of patients | 51.52 [49.02 to 54.01]

2. Secondary Outcome: Changes in the PF-10 Score From Visit 1 to Visit 2
Description: Change in PF-10 score was determined by taking into account the individual change of each patient between Baseline (Visit 1) and Week 6 (approx.) (Visit 2).
Time Frame: baseline and approx. week 6
Population: FAS
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 1578
Unit on Scale | 11.63 (19.04)

3. Secondary Outcome: General Condition of the Patient, Evaluated by the Physician (PGE Score) at Visit 1 and Visit 2.
Description: Physician's Global Evaluation (PGE) score documented by physicians at visit 1 (baseline) and at visit 2 (approx. 6 weeks later). the PGE score documented from 1 to 8. The highest value (=8) representing an excellent general condition
Time Frame: Baseline (Visit 1) and Week 6 (approx.) (Visit 2)
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 1578
Percentage of participants
  Baseline (Visit 1) : PGE score 1 | 1.20
  Baseline (Visit 1) : PGE score 2 | 11.28
  Baseline (Visit 1) : PGE score 3 | 22.69
  Baseline (Visit 1) : PGE score 4 | 30.04
  Baseline (Visit 1) : PGE score 5 | 18.82
  Baseline (Visit 1) : PGE score 6 | 11.91
  Baseline (Visit 1) : PGE score 7 | 3.61
  Baseline (Visit 1) : PGE score 8 | 0.44
  Week 6 (approx.) (Visit 2): Score 1 | 0.25
  Week 6 (approx.) (Visit 2): Score 2 | 3.68
  Week 6 (approx.) (Visit 2): Score 3 | 10.71
  Week 6 (approx.) (Visit 2): Score 4 | 18.12
  Week 6 (approx.) (Visit 2): Score 5 | 28.33
  Week 6 (approx.) (Visit 2): Score 6 | 24.97
  Week 6 (approx.) (Visit 2): Score 7 | 11.98
  Week 6 (approx.) (Visit 2): Score 8 | 1.71
  Week 6 (approx.) (Visit 2): missing | 0.25

4. Secondary Outcome: Patient Overall Satisfaction With Spiolto® Respimat® at Week 6 (Approx.) (Visit 2).
Description: At Week 6 (approx.) (Visit 2) patients were asked how overall satisfied they were with the Spiolto® Respimat® treatment.
Time Frame: Week 6 (approx.) (Visit 2)
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 1578
Percentage of participants
  Very satisfied | 33.59
  Satisfied | 48.86
  Rather satisfied | 8.11
  Neither satisfied nor dissatisfied | 3.99
  Rather dissatisfied | 2.09
  Dissatisfied | 2.66
  Very dissatisfied | 0.63
  Not answered | 0.06

5. Secondary Outcome: Patient Satisfaction With Inhaling From the Respimat® Device at Week 6 (Approx.) (Visit 2).
Description: At Week 6 (approx.) (Visit 2) patients were asked how satisfied they were by inhaling with the Respimat® device.
Time Frame: Week 6 (approx.) (Visit 2)
Measure: Number; unit: percentage of participants
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 1578
percentage of participants
  Very satisfied | 35.17
  Satisfied | 52.34
  Rather satisfied | 6.91
  Neither satisfied nor dissatisfied | 3.49
  Rather dissatisfied | 0.89
  Dissatisfied | 0.76
  Very dissatisfied | 0.32
  Not answered | 0.13

6. Secondary Outcome: Patient Satisfaction With Handling of the Respimat® Inhalation Device at Week 6 (Approx.) (Visit 2).
Description: At Week 6 (approx.) (Visit 2) patients were asked how satisfied they were with handling of the Respimat® inhalation device
Time Frame: Week 6 (approx.) (Visit 2)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 1578
percentage of participants
  Very satisfied | 33.08
  Satisfied | 52.09
  Rather satisfied | 9.82
  Neither satisfied nor dissatisfied | 2.98
  Rather dissatisfied | 0.82
  Dissatisfied | 0.82
  Very dissatisfied | 0.32
  Not answered | 0.06

ADVERSE EVENTS:
Time Frame: From first drug administration until end of study, up to approx 6 weeks.
Arm/Group | Spiolto Respimat
All-Cause Mortality (participants affected / at risk) | 2/1737
Serious Adverse Events (participants affected / at risk) | 3/1737
Other Adverse Events (participants affected / at risk) | 0/1737
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiolto Respimat (N=1737)
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The impact and the interpretation of this Non Interventional Study (NIS) data are limited due to NIS concept

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT02675517/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT02675517/SAP_001.pdf